CLINICAL TRIAL: NCT06273059
Title: Genomic Study of Young-Onset Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dicky L Tahapary, Dr, Indonesia University
Other Study IDs: 22-07-0717
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Genomic; Diabetes Mellitus; MODY
Keywords: Genomic; Diabetes mellitus; MODY
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Subjects will be taken 40 ml of blood sample. Around 30 ml from the blood sample will be used for genomic examination and biobanking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients and Healthy controls: Diabetic patients and Healthy controls

SUMMARY:
Diabetes Mellitus (DM) has been a major contributor to health burden in Indonesia and currently its burden still continues to rise. This is a result of increasing DM prevalence in the country as well as high rates of chronic complications from DM. Findings in Indonesia show that there is a high proportion of young people with diabetes, and also a high risk of therapeutic failure and complications from DM occurring in the younger population.

Young-onset DM has a wide clinical spectrum, including autoimmune DM, polygenic DM, and monogenic DM such as Mature Onset Diabetes of the Young (MODY). Identification and proper diagnosis of young-onset DM spectrum is crucial to treatment outcomes, as certain spectrums, such as some subtypes of MODY, may benefit from cost-efficient alternatives with better outcomes.

However, proper diagnosis of young-onset DM in Indonesia is still a great challenge, as currently some examinations, including genetic testing, has not yet been feasibly done in the country. With current advances in genomics, genetic testing may prove to be fundamental in providing optimal and personalized treatment and care for DM patients.

This study is a pilot project aimed to initiate genomic research in young-onset DM patients in Indonesia. In the short term, this study aims to identify genetic variants that may be able to increase diagnostic accuracy of the young-onset DM spectrum. In the long term, this study aims to identify new genetic variants of young-onset DM. The study also aims to identify genetic variants associated with risks of chronic complications.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a progressive, degenerative chronic disease which clinically manifests as hyperglycemia due to resistance and/or insulin deficiency.(1) According to data from the International Diabetes Federation (IDF), in 2017, around 425 million people in the world have diabetes, and it is predicted that this figure would increase up to 629 million by 2045.(2) Currently, diabetes has become a major contributor to health burden and its prevalence has been steadily increasing. Indonesia places sixth among countries with the highest number of people with diabetes with around 10.3 million in 2017(2) which then increase to more than 19 million in 2021. This is aligned with an increase in diabetes mellitus (DM) prevalence in Indonesia from 5,6% in 2007 to 10,9% in 2018. (3,4) The high prevalence of DM in Indonesia causes great burden in its health sector, both directly and indirectly. Most of the burden brought by DMT2 is contributed by various possible complications as the disease progresses. (1) Chronic complications of DMT2 comprises of vascular disorders, both microangiopathy or macroangiopathy, metabolic disorders and increased risk of infection. (5) Microangiopathy complications include retinopathy which may lead to blindness, nephropathy which may lead to kidney failure, peripheral neuropathy which may severely affect quality of life and diabetic cardiopathy which may lead to heart failure. Macroangiopathy complications include coronary heart disease, stroke, and peripheral artery disease (PAD) which may lead to amputation. (5) Other complications include increased risk of liver cirrhosis due to fatty liver, sexual dysfunction, and increased risk of certain infections such as tuberculosis (TB). (6-8) DM is also associated with higher risk of mortality from COVID-19.

Several studies show that the rate of complications from DM is quite high. According to a study from Dr. Cipto Mangunkusumo National General Hospital in 2011, neuropathy is found to be the most frequent complication (54%), followed by retinopathy (33.4%) and proteinuria (26.5%). (9,10) Two major factors which contribute to these frequent rates of complications are late diagnosis and poor glycemic control. Another finding which may also contribute to this phenomenon is that there is a high proportion of young people with diabetes in Indonesia, whereby studies show that DM in young people has higher risks of therapeutic failure and chronic complications. (11, 12) The high rates of therapeutic failure and chronic complications in people with young-onset DM may greatly affect not only directly through financial burden from healthcare, but also indirectly through arising problems in daily life such as decreased productivity. Diabetics with chronic complication may spend more time in healthcare facilities rather than in other activities, compromising work productivity. Hence, a sufficient understanding of risk factors and clinical spectrums of young-onset DM is important for providing optimal care.

Ethnicity and intrauterine environment might be strong predictors of young-onset T2DM. (11) Obesity, history of low birth weight, and genetic factors also contribute significant roles. (11) The clinical spectrum of young-onset DM varies, including autoimmune DM, polygenic DM, and monogenic DM such as Mature Onset Diabetes of the Young (MODY). Accurate diagnosis plays an important role in providing proper treatment to prevent chronic complications.

MODY is a monogenic form of diabetes in the form of autosomal dominant non-insulin dependent diabetes. (13) MODY contributes to 1-5% of DM cases and symptoms generally appear at a young age (<25 years old). MODY is commonly misdiagnosed as type 1 DM (T1DM) or T2DM. Molecular diagnosis is needed for the accurate diagnosis and optimal treatment of MODY. It also provides possible means to screen and provide early diagnosis of asymptomatic family members. (13) Some subtypes of MODY (HNF1A, HNF4A, KCNJ11, dan ABCC8) may optimally be treated with sulfonylureas, which would be more cost-efficient and provide better clinical outcomes compared to insulin therapy. However, this has not been feasible in Indonesia as some examinations, especially genetic testing, may only be performed by sending samples overseas which would cost greatly. This has proved to be an obstacle to providing tailored or personalized therapy for patients. Personalised medicine involves not only giving accurate diagnosis, but also providing proper choice of therapy as well as predicting possible complications that may appear so that intervention may be done early in their course. To achieve this, genetic testing might be fundamental. In the present, genomic testing in DM is rapidly and continuously developing. This study aims to initiate genomic research in young-onset DM patients in Indonesia. In the short term, this study aims to identify genetic variants that may be able to increase diagnostic accuracy of the young-onset DM spectrum. This may also serve as a baseline for providing personalised medicine care. In the long term, this study aims to identify new genetic variants of young-onset DM.

RESEARCH OBJECTIVES The overall objective of this study is to identify and describe genetic variation of young-onset DM in Indonesia.

The specific objectives are:

1. To describe the proportion of MODY in young-onset DM.
2. To describe genetic variation of MODY in Indonesia.
3. To describe genetic variation in young-onset DM with diabetic complications in various systems:

   1. Cardiovascular complications: coronary heart disease (CHD) and diabetic cardiomyopathy
   2. Peripheral vascular complications
   3. Neurological complications: cerebrovascular disease (CVD) and peripheral neuropathy
   4. Diabetic nephropathy
   5. Diabetic retinopathy
   6. Fatty liver and fatty pancreas
   7. Hearing impairment
   8. Sexual dysfunction

Study Population and Sample The study population is early-onset DM patients. Subjects will be recruited from outpatient clinics Dr. Cipto Mangunkusumo National General Hospital metabolic and endocrine outpatient clinic and KIARA pediatric endocrine outpatient clinic from September 2022 to April 2024. The study will also recruit healthy controls who fulfill the inclusion criteria. Healthy controls will be recruited from Dr. Cipto Mangunkusumo National General Hospital employees undergoing medical checkups and the general population if target sample size has not been met. The study aims to recruit 1,000 diabetic patients and 1,000 healthy controls.

Diabetic patients Inclusion criteria

* Diabetic patient fulfilling criteria from Indonesian Endocrinology Association (PERKENI) 2021 guidelines:

  * Fasting blood glucose 126 mg/dL
  * 2-hour post oral glucose blood glucose/oral glucose tolerance test 200 mg/dL
  * HbA1c 6.5%
  * Random blood glucose 200 mg/dL with classic symptoms or hyperglycemic crisis.
* Patients aged 8-40 years old when diagnosed with diabetes mellitus
* Registered in Dr. Cipto Mangunkusumo National General Hospital and satellite hospitals
* Willing to participate in the study with proof of informed consent agreement Exclusion criteria
* Subject is experiencing severe illness

Healthy controls Inclusion criteria

* Aged 8-40 years old
* Fulfilling criteria of normal blood glucose levels according to Indonesian Endocrinology Association (PERKENI) 2021 guidelines:

  * Fasting blood glucose 100 mg/dL
  * 2-hour post oral glucose blood glucose/oral glucose tolerance test 140 mg/dL
  * HbA1c 5.7% Exclusion criteria
* Subject is unwilling to participate in the study

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients

  * Diabetic patient fulfilling criteria from Indonesian Endocrinology Association (PERKENI) 2021 guidelines:

    * Fasting blood glucose 126 mg/dL
    * 2-hour post oral glucose blood glucose/oral glucose tolerance test 200 mg/dL
    * HbA1c 6.5%
    * Random blood glucose 200 mg/dL with classic symptoms or hyperglycemic crisis.
  * Patients aged 8-40 years old when diagnosed with diabetes mellitus
  * Registered in Dr. Cipto Mangunkusumo National General Hospital and satellite hospitals
  * Willing to participate in the study with proof of informed consent agreement

Exclusion Criteria:

* Subject is experiencing severe illness

Healthy controls Inclusion criteria

* Aged 8-40 years old
* Fulfilling criteria of normal blood glucose levels according to Indonesian Endocrinology Association (PERKENI) 2021 guidelines:

  * Fasting blood glucose 100 mg/dL
  * 2-hour post oral glucose blood glucose/oral glucose tolerance test 140 mg/dL
  * HbA1c 5.7% Exclusion criteria
* Subject is unwilling to participate in the study

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population is early-onset DM patients. Subjects will be recruited from outpatient clinics Dr. Cipto Mangunkusumo National General Hospital metabolic and endocrine outpatient clinic and KIARA pediatric endocrine outpatient clinic from September 2022 to April 2024. The study will also recruit healthy controls who fulfill the inclusion criteria. Healthy controls will be recruited from Dr. Cipto Mangunkusumo National General Hospital employees undergoing medical checkups and the general population if target sample size has not been met. The study aims to recruit 1,000 diabetic patients and 1,000 healthy controls.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
The overall objective of this study is to identify and describe genetic variation of young-onset DM in Indonesia. | 1 years

SECONDARY OUTCOMES:
To describe the proportion of MODY in young-onset DM | 1 years
To describe genetic variation of MODY in Indonesia. | 1 years
To describe genetic variation in young-onset DM with diabetic complications in various systems: | 1 years
  Cardiovascular complications: coronary heart disease (CHD) and diabetic cardiomyopathy b. Peripheral vascular complications c. Neurological complications: cerebrovascular disease (CVD) and peripheral neuropathy d. Diabetic nephropathy e. Diabetic retinopathy f. Fatty liver and fatty pancreas g. Hearing impairment h. Sexual dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Dicky Tahapary, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No